CLINICAL TRIAL: NCT06570226
Title: Discussion on the Effectiveness of Tea on Blood Pressure, Body Composition and Vision Problems in College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Responsible Party: Principal Investigator, Ciao-Lin Ho, Assistant Professor, Hungkuang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLHo
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Myopia; Visual Fatigue; Blood Pressure; Body Composition; Body Fat
Keywords: Roselle tea; myopia; college students; body composition; anthocyanin
MeSH Terms: conditions — Myopia; Asthenopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the hibiscus tea group (Experimental): To drink the hibiscus tea for 10 weeks. At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, the visual fatigue scale, blood pressure, and body composition were examined respectively. At the initial stage (0th week) and at the 10th week after stopping drinking, visual acuity examinations were performed.
  Interventions: Dietary Supplement: hibiscus tea
- the boiled water drinking group (No Intervention): To drink the boiled water for 10 weeks. At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, the visual fatigue scale, blood pressure, and body composition were examined respectively. At the initial stage (0th week) and at the 10th week after stopping drinking, visual acuity examinations were performed.

INTERVENTIONS:
Dietary Supplement: hibiscus tea — Some cell and animal experiments have pointed out that drinking tea may be related to hypotension, body composition and vision problems, and there are more and more related advertisements, especially for hibiscus tea, which is rich in anthocyanins.
  Arms: the hibiscus tea group

SUMMARY:
Background:

Tea is a universal beverage and one of the most popular drinks around the world. Some cell and animal experiments have pointed out that drinking tea may be related to hypotension, body composition and vision problems, and there are more and more related advertisements, especially for hibiscus tea, which is rich in anthocyanins. However, there is a lack of literature on the effectiveness of hibiscus tea drinks in preventing and treating blood pressure, body composition and vision problems in college students.

Purposes:

This study used a randomized human trial to evaluate the effects of drinking hibiscus tea on the control and reduction of blood pressure, body composition, and near vision problems. 100 subjects were divided into 2 groups: the hibiscus tea group and the boiled water drinking group, and they continued to drink it for 10 weeks. At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, the visual fatigue scale, blood pressure, and body composition were examined respectively. At the initial stage (0th week) and at the 10th week after stopping drinking, visual acuity examinations were performed.

Expected results:

1. To explore the effect of hibiscus tea drinks on subjects' myopia.
2. To explore the effect of hibiscus tea drinks on visual fatigue of subjects.
3. To explore the effect of hibiscus tea drinks on the blood pressure of subjects.
4. To explore the impact of hibiscus tea drinks on the body composition of subjects.
5. To explore the effect of hibiscus tea drinks on body fat of subjects.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are college students aged 15 to 22 years old. -

Exclusion Criteria:

* hemodialysis patients who need to limit their water intake
* those with a history of gastric ulcers
* those allergic to anthocyanins
* those who have long-term consumption or consumption of beverages, foods or health products containing high anthocyanins that may interfere with the study after evaluation, for example: foods or health foods such as cranberries, blueberries, cherries and grapes.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
To explore the effect of hibiscus tea drinks on subjects' myopia. | At the beginning of the trial (week zero) and the tenth week
  At the beginning of the trial (week zero), and the tenth week after stopping drinking, Myopia (spherical equivalent refractive error, unit: diopter) was examined.
To explore the effect of hibiscus tea drinks on visual fatigue of subjects. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, the visual fatigue scale was examined by Visual Fatigue Questionnaire (Heuer et al,1989).
  Heuer, H., Hollendiek, G., Kröger, H., & Römer, T. (1989). Rest position of the eyes and its effect on viewing distance and visual fatigue in computer display work. Zeitschrift fur experimentelle und angewandte Psychologie, 36(4), 538-566.
To explore the effect of hibiscus tea drinks on the blood pressure of subjects. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, blood pressure (mmHg) was examined.
To explore the impact of hibiscus tea drinks on weight. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, weight (kg) was examined.
To explore the impact of hibiscus tea drinks on muscle mass for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, muscle mass (kg) was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on muscle quality for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, muscle quality (MQ) was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). MQ = muscle strength (kg)/muscle mass (kg). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on physique ratings for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, physique ratings was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Physique ratings were determined as follows: 1-Hidden Excess Fat, 2-Medium Frame & Excess Fat, 3-Solidly Built, 4-Low Muscle, 5-Standard, 6-Muscular, 7-Low Muscle & Low Fat, 8-Thin & Muscular (Athlete), and 9-Very Muscular (Athlete). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on Visceral Fat for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, Visceral Fat was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Based on all the available information it gives you a range between 1 and 59. A rating between 1 and 12 indicates that you have a healthy level of visceral fat. A rating between 13 and 59 indicates that you have an excessive level of visceral fat.Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on BMR (Basal Metabolic Rate) for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, BMR (kcal) was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page, Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on total body water (%) for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, total body water (%) was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). The ideal percentage for adult women will fluctuate between 45 and 60%, while the ideal percentage for adult men will be between 50 and 65% of the total body. Tanita Home Page, Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on BONE MASS for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, BONE MASS (kg) was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page, Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on BMI for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, BMI (kg/m^2) was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page, Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the impact of hibiscus tea drinks on Metabolic age for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, Metabolic age was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page, Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
To explore the effect of hibiscus tea drinks on body fat percentage of subjects for body composition. | At the beginning of the trial (week zero), the second week, the sixth week and the tenth week
  At the beginning of the trial (week zero), the second week, the sixth week, and the tenth week after stopping drinking, body fat percentage (%) was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). .

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kang Ning, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No